CLINICAL TRIAL: NCT03198949
Title: A Prospective, Randomized, Double-blind, Placebo-controlled Cross Over Study Investigating the Anti-epileptic Efficacy of Afinitor (Everolimus) in Patients With Refractory Seizures Who Have Focal Cortical Dysplasia Type II (FCD II)
Brief Title: A Study Investigating the Anti-epileptic Efficacy of Afinitor (Everolimus) in Patients With Refractory Seizures Who Have Focal Cortical Dysplasia Type II (FCD II)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4-2017-0299
Record Dates: First submitted 2017-06-13; First posted 2017-06-26 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Epilepsy and Focal Cortical Dysplasia II
MeSH Terms: conditions — Epilepsy | interventions — Everolimus

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized, double-blind, placebo-controlled cross over study to evaluate the efficacy and safety of everolimus (trough 5-15 ng/mL) given as adjunctive therapy in patients with FCDII who already failed more than 2 antiepileptic drugs and surgery.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: During baseline phase and core phase, double-blind is maintained. Only one independent investigator who check trough drug level of everolimus and and one pharmacist who dispenses IND will be exposed. All the rest of the researchers will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- everolimus first arm (Experimental): All subjects will receive everolimus during Core phase I and placebo during Core phase II.
  Interventions: Drug: Afinitor (everolimus)
- placebo first arm (Placebo Comparator): All subjects will receive placebo during Core phase I and everolimus during Core phase II.
  Interventions: Drug: Afinitor (everolimus)

INTERVENTIONS:
Drug: Afinitor (everolimus) — Everolimus doses will be 4.5mg/m2 po daily given at first time and then during the 4-week titration period everolimus dose may get adjusted to reach trough concentration of 5 - 15 ng/mL.
  (In order to keep the blind, placebo doses will be also adjusted during core phase based on a random scheme of dose changes.)

SUMMARY:
This is a prospective, randomized, double-blind, placebo-controlled cross over study designed to evaluate the efficacy and safety of everolimus (trough 5-15 ng/mL) given as adjunctive therapy in patients with focal cortical dysplasia type II who already failed more than two antiepileptic drugs and surgery.

This study will assess the impact of everolimus to placebo on seizure frequency in focal cortical dysplasia type II. The number of patients who experience seizure reduction of 50% or more will be counted during last 4 weeks of each core phase.

DETAILED DESCRIPTION:
This is a prospective, randomized, double-blind, placebo-controlled cross over study to evaluate the efficacy and safety of everolimus (trough 5-15 ng/mL) given as adjunctive therapy in patients with FCDII who already failed more than 2 antiepileptic drugs and surgery.

1. Baseline phase (4 weeks, week -4~-1): From Screening Visit (Week -4, V1) to starting titration visit at Week -1 (V2). For baseline seizure frequency calculations, the 4-week prospective period seizure counts will be totaled. Antiepileptic drug use will be assessed, and patients are required to be on a stable dose of AEDs. All patients who meet eligibility criteria will be randomized in a 1:1 ratio to treatment first arm and placebo first arm.
2. Core phase I (12 weeks, week 0~11) 2.1.Titration I period (4 weeks, week 0~3): Everolimus doses will be 4.5mg/m2 po daily given at first time and then during the 4-week titration period everolimus dose may get adjusted to reach trough concentration of 5 - 15 ng/mL. At week 2 (V3), 3 (V4) pre-dose PK blood samples will be taken for potential dose adjustments.

   2.2. Maintenance I period (8 weeks, week 4~11): After the completion of the titration period, the vast majority of patients are expected to continue at their current dose level during the entire 8 week maintenance period. However, the possibility of further titration does still exist, based on the planned pre-dose PK blood samples that will be collected every 4 weeks [week 4(V5) and 8(V6)].
3. Core phase II (12 weeks, week 12~23): After the completion of the core phase I, the everolimus first group will be changed to the placebo and the placebo first group will take everolimus. Dose titration method is same with core phase I.
4. Unblinded extension phase (29 weeks, week 24-52): After approval, all enrolled patients will be offered the opportunity to enter the unblinded extension phase of the study at the end of week 23 and continue everolimus. Everolimus will be provided to every study patient during the extension phase of 29 weeks. During the extension phase Everolimus doses will be titrated based on pre-dose PK blood samples at week 24 (V12), 28 (V13), 40 (V14), seizure frequency and everolimus tolerability. At week 52 (V15), the final analysis which include serum and CSF PK studies will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between the ages of 4 and 40
* Pathologically confirmed Focal Cortical Dysplasia type II (FCDII)
* Refractory seizure in spite of at least 2 antiepileptic drugs (AEDs) and surgery
* Subjects must have experienced at least 3 seizure events per month for two months retrospectively among 3 months prior to the baseline period in spite of using 1 AED or more.
* Must be at least one antiepileptic drug at a stable dose for at least 4 weeks at the start of the 4-week prospective baseline phase, remain on the same regimen throughout the baseline phase.
* VNS and ketogenic diet are allowed. If the patient is using VNS, device stimulator parameters must remain constant throughout the baseline phase. If the patient is on ketogenic diet, the ratio of the diet must remain constant throughout the baseline phase.
* At least 3 seizures throughout the baseline phase.
* Subjects and their legal guardians must have the ability to comprehend the informed consent form and be willing to provide informed consent. For subjects who are too young or unable to comprehend the written consent, a legal guardian who is able to describe and provide an understanding of the informed consent to the subject must sign the consent form on behalf of the subject.

Exclusion Criteria:

* Patients who need hospitalization due to causes not related to FCDII or epilepsy
* Patients who are pregnant or planning on becoming pregnant
* Patients with seizures secondary to causes other than focal cortical dysplasia
* Immunocompromised patients
* Patients who have received prior treatment with a systemic mTOR inhibitor
* Patients who do not follow up last one year
* Patients who do not show EEG abnormalities
* Patients with a history of non-compliance to medical regimens or who are considered potentially unreliable
* Patients with positive HBV Ag
* Patients who receive live vaccination during baseline study
* Patients with a known hypersensitivity to everolimus or other rapamycin-analogues(sirolimus, temsirolimus) or to its excipients
* Patients who have galactose intolerance, Lapp lactase deficiency, glucose-galactose malabsorption, or other genetic problems related to lactose digestion.

Ages: 4 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2018-05-24 (Actual); Primary Completion 2020-09-11 (Actual); Study Completion 2020-09-11 (Actual)

PRIMARY OUTCOMES:
The number of patients who experience seizure reduction of 50% or more | Seizure frequency during the last 4 weeks of core phase
  During last 4 weeks of core phase, to compare the number of patients who experience seizure reduction of 50% or more on trough range (5-15 ng/mL) of everolimus versus placebo in FCD II with drug-resistant epilepsy

SECONDARY OUTCOMES:
seizure-free days | during last 4 weeks of core phase
  To evaluate seizure-free days during double-blind treatment with adjunctive everolimus compared with placebo
reduction in seizure frequency | during last 4 weeks of core phase
  To compare the reduction in seizure frequency on trough range (5-15 ng/mL) of everolimus versus placebo in patients with FCD II
generalized tonic-clonic seizure-free days | during last 4 weeks of core phase
  To evaluate generalized tonic-clonic seizure-free days during double-blind treatment with adjunctive everolimus compared with placebo
reduction in generalized tonic-clonic seizure frequency | during last 4 weeks of core phase
  To compare the reduction in generalized tonic-clonic seizure frequency on trough range (5-15 ng/mL) of everolimus versus placebo in patients with FCD II
number of patients who experience generalized tonic-clonic seizure reduction of 50% or more | during last 4 weeks of core phase
  To compare the number of patients who experience generalized tonic-clonic seizure reduction of 50% or more on trough range (5-15 ng/mL) of everolimus versus placebo in FCD II
level of everolimus in cerebrospinal fluid (CSF) (ng/mL) | One time measurement of everolimus level in CSF (ng/mL) will be performed after 52 weeks
  Measure level of everolimus in cerebrospinal fluid (CSF) (ng/mL) and compare the value with level of everolimus in blood (ng/mL) in relation to the percentage of seizure reduction in patients who agree to perform CSF analysis additionally. We hypothesize that some patients with target blood everolimus level would not respond to everolimus because CSF everolimus level does not proportionally increase. We aim to find differences in CSF everolimus levels between patients who respond well and patients who respond poorly.
level of everolimus in blood (ng/mL) | measurement of everolimus level in blood (ng/mL) will be performed at week 0, 2, 3, 4, 8, 12, 14, 15, 16, 20, 24, 28, 40, and 52
  To measure the level of everolimus in blood (ng/mL) in relation to the percentage of seizure reduction. We hypothesize that some patients would not respond to everolimus because everolimus level does not proportionally increase with increased intake of everolimus.
adverse events related to everolimus use | Every week during core phase through regular study visits or call visits from week 0 to week 24. At 28, 40, and 52 during extension phase
  Every adverse event which occurs during the study will be collected. CTCAE 4.03 guideline will be used. Number of patients who discontinue using everolimus will be collected and the number will be compared to the number of patients who discontinue placebo during the same period. Reasons of early withdrawal will be collected.

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University Healthcare System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim SH, Kang HC, Roh YH, Hahn J, Min KL, Lee SJ, Yang D, Choi HS, Park S, Lee JH, Lee SG, Kim SH, Chang MJ, Kim HD. Efficacy and safety of everolimus for patients with focal cortical dysplasia type 2. Epilepsia Open. 2025 Feb;10(1):243-257. doi: 10.1002/epi4.13104. Epub 2024 Nov 28. PMID 39607729